CLINICAL TRIAL: NCT07013513
Title: Characterising the Physiological Resilience of People With Parkinson's Disease - With Feasibility
Brief Title: Characterising Physiological Resilience in People With Parkinson's Disease
Acronym: ParkEx
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Bethan Phillips, Professor of Translational Physiology, University of Nottingham
Other Study IDs: FMHS 82-0225
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease, elderly, resilience, characterisation, aerobic exercise, feasibility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parkinson's disease (PD) is a condition that affects movement and gets worse over time. It is more common in older adults. People with PD may have symptoms like shaking, stiff muscles, slow movement, and trouble with balance. They may also experience other issues like pain, depression, anxiety, and memory problems, which can make daily life harder.

Physiological resilience is the body's ability to recover or stay strong despite challenges like aging or illness. People with low resilience may struggle to cope with illness, become less active, and have a higher risk of weakness or hospitalization. Since both PD and low resilience are more common in older adults, understanding how PD affects resilience can help improve care.

This study will look at resilience in people with PD by measuring heart, lung, muscle, coordination, memory, and thinking abilities. It will also compare two types of single-session aerobic exercise-cycling and walking on a treadmill-regarding participants' perspectives. Participants will be randomly chosen to do one of these exercises for 40 minutes at a moderate level. Afterward, they will share their thoughts on how enjoyable and comfortable the exercise was and whether they would continue doing it.

Aerobic exercise is often recommended for people with PD, but it is unclear which type is best for people with PD and which type is mostly preferred by participants with PD. The results of this study will help practitioners make better exercise recommendations for people with PD, leading to better symptom management and a higher quality of life.

DETAILED DESCRIPTION:
Parkinson's is a chronic, progressive, neurodegenerative movement disorder. Both genetic and environmental factors may contribute to the development of Parkinson's in an individual. The onset of PD before the age of 50 is rare but does become more common as people age, affecting ~1% of adults over the age of 60 and 4% of those over 85. The most important motor signs of PD are rest tremor, bradykinesia, rigidity and postural instability. Abnormalities in gait, balance, eye movement, posture, speech, and facial expressions are common. Poor balance, gait disturbance, and impaired mobility are among the most important research priorities identified by people living with PD. Furthermore, people with PD frequently experience non-motor symptoms such as pain, anxiety, depression, dementia, and constipation. Collectively, these symptoms lead to deterioration in quality of life, impaired ability to perform activities of daily living, and reduced functional independence, and motor performance.

Physiological resilience refers to the capacity to retain or regain physical function in the presence of diseases or age-related impairments. Poor resilience may raise the likelihood of being vulnerable to stresses, which could lead to negative functional and clinical consequences like a prolonged course of illness/hospitalization, reduced physical activity, an elevated risk of frailty, and even mortality. It is important to assess older populations' physiological resilience (check their readiness levels for potential future stressors). Since the risk of low resilience and prevalence of PD increase with advanced age, there is a relationship between low physiological resilience and PD due to the fact that it can deteriorate the parameters of resilience. Therefore, it is important to explore the characteristics of physiological resilience in PD populations.

This study will explore the characteristics of physiological resilience in terms of muscle strength, muscle mass, neuromuscular function, functional ability, cardiorespiratory fitness, dexterity, and cognition in people with PD.

Moreover, among the several exercise modalities implemented in the rehabilitation of PD symptoms, aerobic exercise is the most frequently employed and it is also a crucial component of the exercise regimen for people with PD according to European and American guidelines, which has been stated as a beneficial tool to promote physiological resilience at all stages of life. However, there is a lack of information in the literature on which aerobic exercise modality is better for this purpose in people with PD. Beyond the investigation of physiological resilience parameters in individuals with PD, this study will also provide valuable feedback from this population group on two single-bout aerobic exercises (cycling vs treadmill walking). Participants will be randomised to conduct either cycling or treadmill walking. Each of these two aerobic exercise sessions will last for 40 minutes and will be conducted at moderate intensity (estimated according to the heart rate maximum (HRmax)). Having conducted a single-bout aerobic exercise session; participants will be asked to complete scales about 'exercise enjoyment, tolerability, emotional state, and intention to continue exercising' as feedback. This study will inform future guidelines for exercise prescriptions for PD rehabilitation. It will be a cross-sectional study that collects data at a single-time point.

Potential participants identified will be sent the PIS. The study will be explained via email or over the phone by a member of the research team if needed. Participants who are willing to participate in the study will then be invited to attend the Medical school at the Royal Derby Hospital site for a screening session. The study will include two visits: 1) screening day, 2) assessment day. We will have a pre-screening via telephone call or email to check they meet the eligibility criteria: diagnosed with PD, adequately mobile (able to walk 30 meters), and willing to take part. If these initial points are satisfied, then participants will be invited for a screening session.

At the screening session, written informed consent will be received from the participants since it is an essential legal and ethical consideration before conducting tests for exercising in health, fitness, and clinical settings. Following completion of the consent process, heart rate, blood pressure, ECG, and medical history including previous and current medication usage will be collected via a screening sheet. The unified Parkinson's disease rating scale (UPDRS) will be used to evaluate the severity of PD. This scale consists of 42 items divided into four categories: Section I (mentation, behaviour, and mood), Section II (activities of daily living, graded as "on" or "off"), Section III (motor exam), and Section IV (complications). The UPDRS battery also includes the Hoehn and Yahr, and the Schwab and England scales.

Participants will have a chance to ask any questions about the study protocol, screening, and eligibility assessments. Screening results will be discussed with a clinician to decide participants' eligibility. If an abnormal screening result is encountered, this will be discussed with the participant, and their GP will be informed in writing. Only those parts of the assessment visit that participants feel comfortable performing will be required of. Participants will have direct supervision from a member of the research team at all times.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are willing and able to give informed consent for participation in the study
* Participants who can walk 30 meters with or without walking aids
* Participants who have a confirmed diagnosis of Parkinson's disease by a healthcare professional.

Exclusion Criteria:

* Cardio- and/or pulmonary diseases except for well-controlled hypertension and asthma
* Severe cognitive impairment/dementia
* Joint disorders preventing exercise participation
* Current or recent (<2 years) malignancy (excluding minor cancers such as skin cancer, or not receiving chemotherapy or radiotherapy within the last 3 months)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected from the community sample at local groups that cater to older persons in general, through our current PPI-E networks, and through nonprofit organisations and charities that assist Parkinson's sufferers. The planned study's benefits, inherent risks, potential adverse events, and anticipated time commitments would all be thoroughly explained to volunteers, along with the methods and protocols that will be used. Interested participants then will be assessed according to the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Body mass assessment | on the assessment day (a single time point)
  Bioelectrical impedance analysis (BIA) will be used for this. BIA is simple to use, places a minimal burden on individuals, uses lightweight and inexpensive equipment, and, most significantly, provides no radiation risk compared to many other methods. It is also found feasible and reliable for the measurement of muscle mass for adults in clinical settings.
Muscle mass assessment | on the assessment day (a single time point)
  Muscle thickness, pennation angle, and fascicle length of vastus lateralis will be measured on ultrasound. Ultrasonography is also a technology that is portable, safe, and clearly distinguishes between muscle and subcutaneous fat tissues as well as a valid and novel tool for muscle mass assessment.
Muscle strength with maximum voluntary contraction of knee extension | on the assessment day (a single time point)
  Maximum voluntary contraction is a standardised technique for assessing muscle strength. Knee extension strength will be measured with an isometric dynamometer.
Handgrip strength assessment | on the assessment day (a single time point)
  Isometric hand grip strength is closely correlated with the strength of the muscles in the lower extremities, the torque of the knee, and poor mobility is clinically indicated by low handgrip strength. Higher values mean better results. It will be assessed with a dynamometer.
Surface Electromyography for vastus lateralis, including neuromuscular tracking tasks for knee extension | on the assessment day (a single time point)
  Muscle contraction is initiated by motor units, which are made up of a motor neuron and the muscle fibers it innervates. When a motor unit fires, it generates a compound action potential composed of the synchronized action potentials of the muscle fibers within that unit. Surface EMG electrodes are placed on the skin and pick up the electrical activity generated by these action potentials, representing the overall muscle activity. Force accuracy is an important parameter since most daily activities are conducted at submaximal levels, where force fluctuation can be observed and reduce the ability to create an intended movement. Participants will be requested to follow a force trace line on a monitor during knee extension. The tasks will be performed at levels relative to the MVC ranging from 10-70% of maximum
Cardiorespiratory fitness assessment via 6-minute walking test (6MWT) | on the assessment day (a single time point)
  In the 6MWT, participants are encouraged to walk as much as they can for six minutes along a continuous, interior track that is 30 metres long and has a hard surface. It is a simple, cost-effective, and validated tool in several populations, and it has been frequently used to measure cardiorespiratory fitness as a field test. The distance covered on this test is reported. Higher values mean better results.
Cardiorespiratory fitness assessment via the Ekblom-bak test | on the assessment day (a single time point)
  The Ekblom-bak test consists of exercise at one standardized, low work rate followed by a higher, individually set work rate. Both work rates are performed for 4 minutes at a cadence of 60rpm on a cycle ergometer. The individual higher work rate is chosen by the researcher according to the participants' gender, age, and training background. The higher work rate aims to reach the Borg RPE 12-16. Heart rate is measured during the last minute of each work rate (at 3:15, 3:30, 3:45, and 4:00). Then VO2max is estimated with a formula.
Different balance tasks and balance time on a motion platform (FootScan) | on the assessment day (a single time point)
  For the balance tests, using a platform (FootScan) that can assess features such as Centre of Pressure (COP) and sway, participants will be asked to stand on both feet and then on one foot with their eyes open and closed. Time to failure (i.e., need to place the second foot on the floor and/or open eyes) will be recorded. A chair will be located behind participants for this assessment and a researcher will remain within touching distance. Participants will only be requested to complete the aspects of this assessment that they feel comfortable doing.
Functional ability assessment via short physical performance battery test | on the assessment day (a single time point)
  Short physical performance battery test (SPPB) includes the chair rise, balance, walk and gait speed assessments for functional mobility (24). An overall score is determined on a scale from 0 to 12, with lower scores representing a more severe level of disability and higher scores representing more functionally normal levels.
Functional ability assessment via the Timed up and Go test | on the assessment day (a single time point)
  The Timed up and Go test is a tool for assessing lower limb functional ability and its use has been recommended by the literature. The time required to finish the test is commonly utilised as the primary outcome of the evaluation. This test has previously been used in several studies to assess functional ability
Gait analysis with a walking sensor | on the assessment day (a single time point)
  For this analysis participants simply have to walk over a biomechanics platform while wearing a walking sensor using their normal gait so that features such as stride length and stride symmetry can be assessed
Cognition assessment via Mini-ACE | on the assessment day (a single time point)
  The Mini-ACE is a brief cognitive test that evaluates four main cognitive areas (orientation, memory, language and visuospatial function). Higher values mean better results.
Hand dexterity assessment via 9-hole peg board task | on the assessment day (a single time point)
  Manual dexterity is an important ability that affects an individual's independence in activities of daily living and should be measured as a core element. The 9-hole peg test has been shown to be a valid and reliable tool to measure upper extremity dexterity in various groups

SECONDARY OUTCOMES:
Enjoyment via the Physical Activity Enjoyment Scale on a single-bout aerobic exercise session (either treadmill or cycling) | on the assessment day (a single time point)
  The Physical Activity Enjoyment Scale (PACES) is a questionnaire used to measure the extent to which individuals enjoy engaging in physical activity. It's a tool for understanding the positive emotional experience associated with exercise, which can be a key factor in promoting long-term adherence to physical activity programs. Responses will be indicated indicated on a Likert scale with 18-item version, with higher scores representing greater enjoyment.
Tolerability via the Visual Analog Scale | on the assessment day (a single time point)
  The Visual Analog Scale (VAS) is a method for measuring the intensity of a subjective experience, like pain or discomfort, by having individuals mark a line to indicate their level. It is a continuous scale, typically from 0 to 100, where 0 represents "no pain" and 100 represents "worst possible pain". Tolerability, in this context, often refers to how well a patient can bear a treatment or condition based on the VAS score.
Emotional state assessment via the Feeling Scale | on the assessment day (a single time point)
  The Feeling Scale (FS) is used to measure the emotional state during an exercise session by assessing the pleasure or displeasure experienced by the individual. It is an 11-point bipolar scale ranging from -5 (very bad) to +5 (very good), with verbal anchors like "very bad," "bad," "fairly bad," "neutral," "fairly good," "good," and "very good".
intention to continue exercising assessment via a 7-point Likert scale | on the assessment day (a single time point)
  A 7-point Likert scale can be used to assess intention to continue exercising by asking individuals to rate their agreement with statements like "I plan to continue exercising in the next week" or "I am determined to make exercise a regular part of my life."

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet C Yildirim, Study Director — The University of Nottingham
Locations (1):
- The University of Nottingham/Medical School, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang YC, Bohannon RW, Kapellusch J, Garg A, Gershon RC. Dexterity as measured with the 9-Hole Peg Test (9-HPT) across the age span. J Hand Ther. 2015 Jan-Mar;28(1):53-9; quiz 60. doi: 10.1016/j.jht.2014.09.002. Epub 2014 Sep 28. PMID 25449717
- [Background] Singh NB, Arampatzis A, Duda G, Heller MO, Taylor WR. Effect of fatigue on force fluctuations in knee extensors in young adults. Philos Trans A Math Phys Eng Sci. 2010 Jun 13;368(1920):2783-98. doi: 10.1098/rsta.2010.0091. PMID 20439273
- [Background] Santana MG, de Lira CA, Passos GS, Santos CA, Silva AH, Yoshida CH, Tufik S, de Mello MT. Is the six-minute walk test appropriate for detecting changes in cardiorespiratory fitness in healthy elderly men? J Sci Med Sport. 2012 May;15(3):259-65. doi: 10.1016/j.jsams.2011.11.249. Epub 2011 Dec 11. PMID 22154397
- [Background] Dourado VZ, Nishiaka RK, Simoes MSMP, Lauria VT, Tanni SE, Godoy I, Gagliardi ART, Romiti M, Arantes RL. Classification of cardiorespiratory fitness using the six-minute walk test in adults: Comparison with cardiopulmonary exercise testing. Pulmonology. 2021 Nov-Dec;27(6):500-508. doi: 10.1016/j.pulmoe.2021.03.006. Epub 2021 May 4. PMID 33958319
- [Background] Przkora R, Kinsky MP, Fisher SR, Babl C, Heyde CE, Vasilopoulos T, Kaye AD, Volpi E. Functional Improvements Utilizing the Short Physical Performance Battery (SPPB) in the Elderly after Epidural Steroid Injections. Curr Pain Headache Rep. 2019 Feb 22;23(2):14. doi: 10.1007/s11916-019-0748-2. PMID 30796532
- [Background] Gojanovic M, Holloway-Kew KL, Hyde NK, Mohebbi M, Shivappa N, Hebert JR, O'Neil A, Pasco JA. The Dietary Inflammatory Index Is Associated with Low Muscle Mass and Low Muscle Function in Older Australians. Nutrients. 2021 Apr 1;13(4):1166. doi: 10.3390/nu13041166. PMID 33916033
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Lauretani F, Russo CR, Bandinelli S, Bartali B, Cavazzini C, Di Iorio A, Corsi AM, Rantanen T, Guralnik JM, Ferrucci L. Age-associated changes in skeletal muscles and their effect on mobility: an operational diagnosis of sarcopenia. J Appl Physiol (1985). 2003 Nov;95(5):1851-60. doi: 10.1152/japplphysiol.00246.2003. PMID 14555665
- [Background] Meldrum D, Cahalane E, Conroy R, Fitzgerald D, Hardiman O. Maximum voluntary isometric contraction: reference values and clinical application. Amyotroph Lateral Scler. 2007 Feb;8(1):47-55. doi: 10.1080/17482960601012491. PMID 17364436
- [Background] Scott JM, Martin DS, Ploutz-Snyder R, Matz T, Caine T, Downs M, Hackney K, Buxton R, Ryder JW, Ploutz-Snyder L. Panoramic ultrasound: a novel and valid tool for monitoring change in muscle mass. J Cachexia Sarcopenia Muscle. 2017 Jun;8(3):475-481. doi: 10.1002/jcsm.12172. Epub 2017 Jan 3. PMID 28052593
- [Background] Mijnarends DM, Meijers JM, Halfens RJ, ter Borg S, Luiking YC, Verlaan S, Schoberer D, Cruz Jentoft AJ, van Loon LJ, Schols JM. Validity and reliability of tools to measure muscle mass, strength, and physical performance in community-dwelling older people: a systematic review. J Am Med Dir Assoc. 2013 Mar;14(3):170-8. doi: 10.1016/j.jamda.2012.10.009. Epub 2012 Dec 29. PMID 23276432
- [Background] Lee SY, Ahn S, Kim YJ, Ji MJ, Kim KM, Choi SH, Jang HC, Lim S. Comparison between Dual-Energy X-ray Absorptiometry and Bioelectrical Impedance Analyses for Accuracy in Measuring Whole Body Muscle Mass and Appendicular Skeletal Muscle Mass. Nutrients. 2018 Jun 7;10(6):738. doi: 10.3390/nu10060738. PMID 29880741
- [Background] Bjorkman F, Ekblom-Bak E, Ekblom O, Ekblom B. Validity of the revised Ekblom Bak cycle ergometer test in adults. Eur J Appl Physiol. 2016 Sep;116(9):1627-38. doi: 10.1007/s00421-016-3412-0. Epub 2016 Jun 16. PMID 27311582
- [Background] Sampedro-Piquero P, Moreno-Fernandez RD. Building Resilience with Aerobic Exercise: Role of FKBP5. Curr Neuropharmacol. 2021;19(8):1156-1160. doi: 10.2174/1570159X19666210408124937. PMID 33829973
- [Background] Cosco TD, Howse K, Brayne C. Healthy ageing, resilience and wellbeing. Epidemiol Psychiatr Sci. 2017 Dec;26(6):579-583. doi: 10.1017/S2045796017000324. Epub 2017 Jul 6. PMID 28679453
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468
- [Background] Berganzo K, Tijero B, Gonzalez-Eizaguirre A, Somme J, Lezcano E, Gabilondo I, Fernandez M, Zarranz JJ, Gomez-Esteban JC. Motor and non-motor symptoms of Parkinson's disease and their impact on quality of life and on different clinical subgroups. Neurologia. 2016 Nov-Dec;31(9):585-591. doi: 10.1016/j.nrl.2014.10.010. Epub 2014 Dec 17. English, Spanish. PMID 25529173
- [Background] Schapira AHV, Chaudhuri KR, Jenner P. Non-motor features of Parkinson disease. Nat Rev Neurosci. 2017 Jul;18(7):435-450. doi: 10.1038/nrn.2017.62. Epub 2017 Jun 8. PMID 28592904
- [Background] Pan-Montojo F, Anichtchik O, Dening Y, Knels L, Pursche S, Jung R, Jackson S, Gille G, Spillantini MG, Reichmann H, Funk RH. Progression of Parkinson's disease pathology is reproduced by intragastric administration of rotenone in mice. PLoS One. 2010 Jan 19;5(1):e8762. doi: 10.1371/journal.pone.0008762. PMID 20098733
- [Background] Jankovic J. Parkinson's disease: clinical features and diagnosis. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):368-76. doi: 10.1136/jnnp.2007.131045. PMID 18344392
- [Background] Pringsheim T, Jette N, Frolkis A, Steeves TD. The prevalence of Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2014 Nov;29(13):1583-90. doi: 10.1002/mds.25945. Epub 2014 Jun 28. PMID 24976103
- [Background] Alves G, Forsaa EB, Pedersen KF, Dreetz Gjerstad M, Larsen JP. Epidemiology of Parkinson's disease. J Neurol. 2008 Sep;255 Suppl 5:18-32. doi: 10.1007/s00415-008-5004-3. PMID 18787879
- [Background] Kalia LV, Lang AE. Parkinson disease in 2015: Evolving basic, pathological and clinical concepts in PD. Nat Rev Neurol. 2016 Feb;12(2):65-6. doi: 10.1038/nrneurol.2015.249. Epub 2016 Jan 18. No abstract available. PMID 26782330
- See also: Related Info — https://www.parkinsonnet.nl/app/uploads/sites/3/2019/11/eu_guideline_parkinson_guideline_for_pt_s1.pdf